CLINICAL TRIAL: NCT03415152
Title: A Prospective Observational Program Using Digital Technology Tools to Enhance Patient Adherence to Omacor Therapy
Acronym: DIAPAsOn
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: PUFA5004
Record Dates: First submitted 2018-01-03; First posted 2018-01-30 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: History of Myocardial Infarction; Hypertriglyceridemia
Keywords: Omacor; Omega-3-acid ethyl esters; patient adherence; patient reported outcomes
MeSH Terms: conditions — Hypertriglyceridemia; Patient Compliance | interventions — Omacor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Omacor (Omega-3-acid ethyl esters): Adult patients with history of myocardial infarction not earlier than 6 months ago and/or with diagnosis of hypertriglyceridemia who having been prescribed Omacor for at least 6 months.
  Interventions: Drug: Omacor (Omega-3-acid ethyl esters)

INTERVENTIONS:
Drug: Omacor (Omega-3-acid ethyl esters) — Observational study without intervention, Omacor is prescribed in routine manner in accordance with clinical practice and the valid Instruction for Medical Use regarding the dose, duration of therapy, patient population, and therapeutic indication.

SUMMARY:
A prospective observational program using digital technology tools to enhance patient adherence to Omacor therapy

DETAILED DESCRIPTION:
It is known that only 50% of patients with chronic diseases adhere to medical recommendations; at the same time, high patient adherence significantly improve the survival of patients with chronic diseases. The treatment duration required to achieve a significant reduction in the risk of cardiovascular complications is the subject of discussion, but studies demonstrate that long-term therapy for 5 years or more gives the greatest effect. Today, during the era of technological progress, there is a possibility to freely apply information and telecommunication technologies (e.g. cell phones, computer) in different fields, including medicine. Remote monitoring of patients by means of phone calls using structured questionnaires can also significantly improve clinical outcomes (mortality and cardiovascular hospitalizations) by 38%. Unfortunately, in the case of a long-term, usually lifetime, treatment, the use of such methods is still very limited on a large scale.

This prospective observational program will help to explore the use of digital technologies and evaluate their effectiveness to increase patient adherence using an example of patients whose treatment scheme includes Omacor. Physicians and patients will be granted a personal access to the electronic data capture system. The physician will enter data about patients who signed the informed consent into the electronic system. At Visit 1 the patient will be given a card providing the personal access to his/her account in the electronic system. In addition to visits to the physician, the program specifies remote completion of the electronic form by the patient. Additional objective of the program includes raising patients' awareness about the disease due to familiarization with educational materials available in patient personal account in the electronic system.

This study is a prospective observational program within the frames of which Omacor (Omega-3 triglycerides [EPA/docosahexaenoic acid (DHA) = 1.2/1 - 90%]) is prescribed to patients with a history of myocardial infarction within a routine procedure as a part of the combination therapy (in combination with statins, antiaggregants, beta-blockers, angiotensin-converting enzyme inhibitors (ACE)) and/or to patients with hypertriglyceridemia. The population of observed patients will be limited to those who were prescribed Omacor for the first time or not earlier than 3 months after the last dose of Omacor and course of administration is at least 6 months. Discontinuation of the drug product administration by the patient is not the reason for exclusion of the patient from the study. For outcome measures which are applicable, further analysis will be performed in subgroups of patients with the different medication adherence rate: <0,5, 0,5-0,7, ≥0,8 at Visit 2 and Visit 3. Adherence rate will be calculated as the sum of days when patient taken the full prescribed dose of Omacor in period divided by the number of days in period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Patients with history of myocardial infarction not earlier than 6 months ago. AND/OR Patients with diagnosis of hypertriglyceridemia
* Patients having been prescribed Omacor (Omega-3 triglycerides [EPA/DHA = 1.2/1 - 90%]) for at least 6 months AND who have been taking Omacor no more than 14 days at the time of enrollment into the program.
* Patients who can, in the opinion of the Investigator, himself or through immediate relatives's help complete electronic system of data collection through mobile application or web-browser
* Patients who have signed the consent to participate in this program before entering their data in the electronic Case Report Form (eCRF) and who understand their right to discontinue the program at any time

Exclusion Criteria:

* Patients taken medicines (except for Omacor) or nutrition supplements containing omega-3 in any proportions at the time of enrollment into the program OR it has been less than 3 months since last dose of medicines or nutrition supplements containing omega-3 taken.
* Female patients during pregnancy or breastfeeding
* Patients with increased sensitivity to the active substance, excipients, and soy
* Patients with exogenous hypertriglyceridemia (type I hyperchylomicronemia)
* Participation in any other clinical or non-clinical study/program at present or within the latest 30 days
* Patients with any other clinical states that make him/her ineligible for the program on the study doctor's opinion based on clinical assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with myocardial infarction in anamnesis and/or diagnosis of hypertriglyceridemia who are under medical supervision in healthcare institutions of Russia and receive Omacor
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- Russia (93):
  - Gbuz Amokb Jsc, Astrakhan
  - polyclinic GKB №21, Bashkortostan
  - GAUZ "BKDTs", Bryansk
  - GP # 1, Chelyabinsk
  - GKB №3, Chelyabinsk
  - Federal State Budgetary Institution "Research Institute of Complex Problems of Cardiovascular Diseases", Kemerovo
  - GBUZ Polyclinic of City Clinical Hospital № 10, Khabarovsk
  - GP #2, Krasnodar
  - MBUZ GP number 11, Krasnodar
  - Gbuz Kkb #2, Krasnodar
  - GBUZ Regional clinical hospital № 2, Krasnodar
  - Yablonovskaya polyclinic, Krasnodar
  - KKB #1, Krasnodar
  - City Polyclinic №27, Krasnodar
  - GP №27, Krasnodar
  - Llc "Auris", Krasnodar
  - City Polyclinic №7, Krasnodar
  - Clinic Mamme, Krasnodar
  - GP №15, Krasnodar
  - GP №17, Krasnodar
  - Mbuz Gp #17, Krasnodar
  - Gbuz Nii Kkb №1, Krasnodar
  - Gbuz "Nii-Kkb №1", Krasnodar
  - GP №25, Krasnodar
  - MBUZ City Polyclinic #11, Krasnodar
  - Municipal budgetary health institution "City Polyclinic # 11", Krasnodar
  - Mbuz Gkb №1, Krasnodar
  - MC Ultramed, Krasnodar
  - MUZ Polyclinic TsRB Poltava, Krasnodar
  - Medical Center "Modern Cardiology", Krasnodar
  - Clinic "Medicine for All", Krasnodar
  - Policlinic № 1, Krasnoyarsk
  - Maikop City Polyclinic №1, Maykop
  - Polyclinic №52 branch №1, Moscow
  - ГП № 210 branch 2, Moscow
  - FGBU Federal Clinical Research Centre of Russia's Federal Medical-Biological Agency, Moscow
  - Gbuz "Gp #22 Dzm", Moscow
  - Fsbi Enc Mz Rf, Moscow
  - City polyclinic № 22, Moscow
  - GP number 176, Moscow
  - Diagnostic Clinical Center №1, Moscow
  - OOO "Lechebnii center", Moscow
  - City polyclinic № 195, Moscow
  - Outpatient center of CDC #4, Moscow
  - GP №45, Moscow
  - GBUZ City polyclinic # 43 DZM filial #3, Moscow
  - GP №219 branch №4, Moscow
  - Branch №1 DGP #94, Moscow
  - MSU #169, Moscow
  - Medical Center "Health", Moscow
  - Noginsk Central District Hospital, Moscow
  - Hospital SCC RAS in Chernogolovka, Moscow
  - Polyclinic of the National Science Center of the Russian Academy of Sciences in Chernogolovka, Moscow
  - GBUZ NO Pavlovsk CRH, Nizhny Novgorod
  - Llc "Healthy Little Healer", Nizhny Novgorod
  - MC "Sadko", Nizhny Novgorod
  - MC Sadko, Nizhny Novgorod
  - MC Dobrii doctor, Nizhny Novgorod
  - Cst on St.Nizhny Novgorod Oao Rzd, Nizhny Novgorod
  - Polyclinic №7 branch 2, Nizhny Novgorod
  - GP #2, Nizhny Novgorod
  - Gauz Nso Gkp #1, Novosibirsk
  - City Polyclinic № 2, Omsk
  - BUZOO "GP number 12", Omsk
  - Consultative clinic, Regional clinical hospital #2 Rostov region, Rostov
  - GP №16, Rostov
  - Polyclinic GB №7, Rostov
  - NUZ Road Clinical Hospital at the station Rostov-Glavnii JSC "Russian Railways", Rostov
  - MBUZ CRB Myasnitskogo region, Rostov-on-Don
  - Gbou Vpo Pspbgmu Im. I.P. Pavlova Ministry of Health of Russia, Saint Petersburg
  - Fsbi "Szfmits Im. Va Almazova" Ministry of Health of Russia, Saint Petersburg
  - GP №121, Saint Petersburg
  - Non-State Healthcare Institution "Road Clinical Hospital at Samara Station JSC "Russian Railways", Samara
  - Gbuz Sb Sgb #10, Samara
  - GBUZ SO "Samara City Hospital 6", Samara
  - Gbuz Co "Volga Crh", Samara
  - Medical Center on Tupolev, Samara
  - Zhigulevskaya polyclinic, Samara
  - City polyclinic № 2, Saratov
  - OGBUZ Polyclinic №3, Smolensk
  - Gbuz Sk Skkkd, Stavropol
  - Regional Clinical Cardiology Dispensary, Stavropol
  - GBUZ SK "Pyatigorsk GKB № 2", Stavropol
  - Gaus Mkdts, Tatarstan
  - GUZ Citi hospital №13, Tula
  - Guz Gb №13, Tula
  - TOKB KDC, Tula
  - First Cardiac Clinic, Tyumen
  - GBUZ RB Polyclinic № 46, Ufa
  - GBUZ IN city Polyclinic №1, Vladimir
  - Guz "Polyclinic № 5", Volgograd
  - Volgograd Regional Clinical Cardiology Center, Volgograd
  - BUZ IN "Voronezh city clinical polyclinic #7", Voronezh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arutyunov GP, Arutyunov AG, Ageev FT, Fofanova TV. Use of Digital Technology Tools to Characterize Adherence to Prescription-Grade Omega-3 Polyunsaturated Fatty Acid Therapy in Postmyocardial or Hypertriglyceridemic Patients in the DIAPAsOn Study: Prospective Observational Study. JMIR Cardio. 2022 Jul 25;6(2):e37490. doi: 10.2196/37490. PMID 35877173

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Started | 3000
Completed | 1975
Not Completed | 1025

BASELINE CHARACTERISTICS:
Population: A total of 3000 patients signed informed consent and were included in the program. Data of Visit 1 were available for 2572 (85.7%) patients, 1975 patients (65.8% of all who signed informed consent) completed the program per protocol.
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2572
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1600
  >=65 years | 972
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1182
  Male | 1390
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 48
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2518
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Russia | 2572

OUTCOME MEASURES:

1. Primary Outcome: Mean Adherence Rate at the End of the Study (Visit 3)
Description: Mean adherence rate is a ratio of the sum of days when the patient took the full prescribed dose of Omacor in the specified period to the number of days in the period.
Time Frame: 6 months
Population: Population of patients registered in electronic system and reported Omacor administration
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 180
proportion of days | 0.37 (0.38)

2. Secondary Outcome: Mean Score of National Questionnaire of Treatment Compliance (Edited by Fofanova T.V. et al.) at the End of the Study (Visit 3)
Description: The average score for the National questionnaire on therapy compliance for all study duration Visit 1 - Visit 3.
  The text of the National questionnaire of treatment compliance consists of five statements with four options for choice. The answer corresponding to very high compliance is estimated at 3 points, the answer corresponding to high compliance is estimated at 2 points, medium compliance - at 1 point and low compliance - 0 points. The patient can get a maximum of 15 points, a minimum of 0 points. Higher scores mean higher compliance
Time Frame: 6 months
Population: Population of patients attended at Visit 3 (month 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Omacor (Omega-3-acid Ethyl Esters): Adult patients with history of myocardial infarction not earlier than 6 months ago and/or with diagnosis of hypertriglyceridemia who have been prescribed Omacor for at least 6 months.
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 1975
score on a scale | 12.9 (2.99)

3. Secondary Outcome: The Percentage of Patients Who Have Chosen Each of the Suggested Reasons for Therapy Termination
Description: The percentage of patients (%) who have chosen each of the suggested reason for therapy termination.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2572
percentage of participants
  Adverse drug reactions | 0
  Lack of efficacy | 0.08
  Inconvenience of use | 0.43
  Absence at the pharmacy | 0.23
  Other reason | 1.94
  Total | 2.68

4. Secondary Outcome: The Average Score on Each of 8 Scales of Short Form Survey (SF)-36 Quality of Life Questionnaire at Visit 2 and Visit 3 vs. the Baseline (Visit 1)
Description: Mean difference of the average score on each of 8 scales of Short Form Survey (SF)-36 quality of life questionnaire at Visit 2 and Visit 3 versus the baseline.
  36-Item Short Form Survey (SF-36) taps eight health concepts. Each of 36 items is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively, so that a high score defines a more favorable health state.
Time Frame: 3 months, 6 months
Population: Population of patients registered in electronic system and reported Omacor administration
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Omacor (Omega-3-acid Ethyl Esters): Adult patients with history of myocardial infarction not earlier than 6 months ago and/or with diagnosis of hypertriglyceridemia who have been prescribed Omacor for at least 6 months Visit 2 - Visit 1 (3 months)
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 180
score on a scale
  Physical functioning (V2-V1,3 m) | 7.63 (13.4)
  Role limitations due to physical health (V2-V1,3m) | 32.86 (48.42)
  Role limitations due to emotional problems (V2-V1, | 25.71 (32.42)
  Energy/fatique (V2-V1,3m) | 20.81 (14.12)
  Emotional wellbeing (V2-V1,3m) | 22.66 (14.69)
  Social functioning (V2-V1,3m) | 26.43 (25.68)
  Pain (V2-V1,3m) | 8.43 (14.12)
  General health (V2-V1,3m) | -6.14 (10.22)
  Physical functioning (V3-V1,6m) | 6.69 (10.08)
  Role limitations due to physical health (V3-V1,6m) | 29.55 (43.39)
  Role limitations due to emotional problems (V3-V1, | 18.18 (30.39)
  Energy/fatique (V3-V1,6m) | 18.18 (13.59)
  Emotional wellbeing (V3-V1,6m) | 25 (14.56)
  Social functioning (V3-V1,6m) | 16.48 (25.41)
  Pain (V3-V1,6m) | 0.11 (0.53)
  General Health (V3-V1,6m) | -9.83 (12.08)

5. Secondary Outcome: Change of Lipid Profile Parameters at Visit 2 and Visit 3 vs. the Baseline (Visit 1)
Description: Mean difference of lipid profile parameters at Visit 2 and Visit 3 vs. the Baseline (Visit
  1)
Time Frame: 3 months, 6 months
Population: Per protocol population: patients who attended at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2167
mmol/L
  total serum cholesterol (TSC) (V2-V1,3m) | -1 (1.09)
  triglycerides (TG) (V2-V1,3m) | -0.98 (1)
  low-density lipoproteins (LDLP) (V2-V1,3m) | -0.77 (0.92)
  high-density lipoproteins (HDLP) (V2-V1,3m) | 0.15 (0.45)
  total serum cholesterol (TSC) (V3-V1,6m) | -1.32 (1.28)
  triglycerides (TG) (V3-V1,6m) | -1.32 (1.15)
  low-density lipoproteins (LDLP) (V3-V1,6m) | -1.02 (1.02)
  high-density lipoproteins (HDLP) (V3-V1,6m) | 0.2 (0.53)

6. Secondary Outcome: Number of Hospitalizations Due to Cardio-vascular Reasons During 6 Months of the Program
Description: Percentage of patients with hospitalizations due to cardiovascular disease
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2572
percentage of participants
  The presence of hospitalizations | 0.74
  The absence of hospitalizations | 99.26

7. Secondary Outcome: Number of New Cases of Stenocardia During 6 Months of the Program
Description: Percentage of patients with new cases of stenocardia
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2572
percentage of participants
  The presence of new cases of angina pectoris | 0.97
  The absence of new cases of angina pectoris | 99.03

8. Secondary Outcome: Number of Non-fatal Myocardial Infarction Cases During 6 Months of the Program
Description: Percentage of patients with non-fatal myocardial infarction cases
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2572
percentage of participants
  Presence of cases of non-fatal myocardial infarcti | 0.04
  Absence of cases of nonfatal myocardial infarctio | 99.96

9. Secondary Outcome: Number of Cases of Cardio-vascular Death During 6 Months of the Program
Description: Percentage of patients dead due to cardio-vascular death
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2572
percentage of participants | 0.04

10. Secondary Outcome: Mean Adherence Rate at Visit 2
Description: as for outcome 1
Time Frame: 3 months
Population: Population of patients registered in electronic system and reported Omacor administration
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 180
proportion of days | 0.48 (0.4)

11. Secondary Outcome: Change of Mean Adherence Rate by End of the Study (Visit 3) Versus Visit 2
Description: as for outcome 1
Time Frame: 3 months, 6 months
Population: Population of patients registered in electronic system and reported Omacor administration
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 180
proportion of days | 0.24 (0.4)

12. Secondary Outcome: The Percentage of Patients With Adherence Rate <0,5, 0,5-0,7, ≥0,8 at Visit 2 and Visit 3
Description: The percentage of patients with adherence rate <0,5, 0,5-0,7, ≥0,8 at Visit 2 and Visit 3
Time Frame: 3 months, 6 months
Population: Population of patients registered in electronic system and reported Omacor administration
Measure: Number; unit: percentage of participants
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 180
percentage of participants
  Low (<0.5) (V2, 3 m) | 50
  Moderate (0.5 - 0.7) (V2, 3 m) | 15.56
  High (≥0.8) (V2, 3 m) | 34.44
  Low (<0.5) (V3, 6 m) | 75
  Moderate (0.5 - 0.7) (V3, 6 m) | 4.44
  High (≥0.8) (V3, 6 m) | 20.56

13. Secondary Outcome: Mean Score of National Questionnaire of Treatment Compliance (Edited by Fofanova T.V. et al.) [9] at Visit 1, Visit 2
Description: The average score for the National questionnaire on therapy compliance at Visit 1, Visit 2.
  The text of the National questionnaire of treatment compliance consists of five statements with four options for choice. The answer corresponding to very high compliance is estimated at 3 points, the answer corresponding to high compliance is estimated at 2 points, medium compliance - at 1 point and low compliance - 0 points. The patient can get a maximum of 15 points, a minimum of 0 points. Higher scores mean higher compliance
Time Frame: 0 months, 3 months
Population: Per protocol population: patients who attended at least one follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2167
score on a scale
  Mean score (V 1, 0 m) | 12.55 (3.11)
  Mean score (V 2, 3 m) | 12.99 (2.88)

14. Secondary Outcome: Change of Mean Score of National Questionnaire of Treatment Compliance (Edited by Fofanova T.V. et al.) [9] at Visit 2 and Visit 3 Versus Baseline (Visit 1)
Description: The text of the National questionnaire of treatment compliance consists of five statements with four options for choice. The answer corresponding to very high compliance is estimated at 3 points, the answer corresponding to high compliance is estimated at 2 points, medium compliance - at 1 point and low compliance - 0 points. The patient can get a maximum of 15 points, a minimum of 0 points.
  Higher scores mean higher compliance
Time Frame: Baseline, 3 Months, 6 Months
Population: Per protocol population: patients who attended at least one follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
Number analyzed (Participants) | 2167
score on a scale
  Mean difference (V 2-V 1, 3 m) | 0.47 (2.46)
  Mean difference (V 3-V 1, 6 m) | 0.44 (2.52)

ADVERSE EVENTS:
Time Frame: 6 months Adverse drug reactions, serious adverse drug reactions and other safety-related information are reported to sponsor from the inclusion of the patient in the program during Visit 1 until Visit 3.
Description: Adverse drug reactions (ADR) but not adverse events (AE) were collected within the study. In the case of an ADR/SADR or other safety-related data, a physician must notify the sponsor contact person within 24 hours after getting acquainted with this information.
Groups:
- Omacor (Omega-3-acid Ethyl Esters): Adult patients who signed informed consent and were included in the program with history of myocardial infarction not earlier than 6 months ago and/or with diagnosis of hypertriglyceridemia and who have been prescribed Omacor for at least 6 months.
Arm/Group | Omacor (Omega-3-acid Ethyl Esters)
All-Cause Mortality (participants affected / at risk) | 4/3000
Serious Adverse Events (participants affected / at risk) | 0/3000
Other Adverse Events (participants affected / at risk) | 4/3000
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacor (Omega-3-acid Ethyl Esters) (N=3000)
Eructation (Gastrointestinal disorders) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Score on the "G. Health" of the SF-36 scale should not be taken into account due to a technical error occurred at the stage of transferring the scale to the electronic case report form and which affected the results, changing the patient's responses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03415152/Prot_SAP_000.pdf